CLINICAL TRIAL: NCT03681236
Title: The Effect of Alveolar Recruitment Maneuver on Postoperative Pulmonary Complications in Laparoscopic Surgery
Brief Title: The Effect of Alveolar Recruitment Maneuver in Laparoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, LEE YEA JI, Assistant professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: B1708-415-302
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Postoperative Pulmonary Complication
Keywords: Alveolar recruitment, laparoscopic surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No alveolar recruitment maneuver (No Intervention): Applying ventilation with tidal volume 6-8mL/kg (ideal body weight) and PEEP 5cmH₂O
- Alveolar recruitment maneuver (Active Comparator): Applying ventilation with tidal volume 6-8mL/kg (ideal body weight) and PEEP 5cmH₂O. In addition to this, performing alveolar recruitment maneuver at 2 moments: before surgical incision, end of pneumoperitoneum
  Interventions: Procedure: Alveolar recruitment maneuver

INTERVENTIONS:
Procedure: Alveolar recruitment maneuver — Applying plateau pressure 30cmH₂O for 30 seconds to achieve alveolar inflation
  Arms: Alveolar recruitment maneuver

SUMMARY:
Investigating the effect of alveolar recruitment on the incidence of postoperative pulmonary complication in patients who undergo laparoscopic surgery

DETAILED DESCRIPTION:
Comparing ventilation with PEEP (positive end expiratory pressure) to ventilation with PEEP and alveolar recruitment, we expect that alveolar recruitment will reduce the incidence of pulmonary complication in patients undergo laparoscopic surgery. Ventilation with only PEEP is generally not enough to reduce postoperative pulmonary complication effectively.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, ASA I-II, scheduled to elective laparoscopic surgery

Exclusion Criteria:

* Chronic lung disease
* Cardiovascular disease
* ASA class ≥ III
* Receiving ventilation therapy or received within 6 months
* Refusal of participation in study or failure in informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2018-10-04 (Actual); Primary Completion 2023-10-04 (Estimated); Study Completion 2023-12-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative pulmonary complication | Immediately after entering PACU
  Performing lung ultrasound to evaluate if pulmonary complication is occurred

CONTACTS AND LOCATIONS:
Overall Officials: Ah Young Oh, M.D., Ph. D, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, department of Anesthesia and pain, Seongnam, Gyenggo-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bae YK, Nam SW, Oh AY, Kim BY, Koo BW, Han J, Yim S. Effect of the alveolar recruitment maneuver during laparoscopic colorectal surgery on postoperative pulmonary complications: A randomized controlled trial. PLoS One. 2024 May 9;19(5):e0302884. doi: 10.1371/journal.pone.0302884. eCollection 2024. PMID 38722838